CLINICAL TRIAL: NCT01012050
Title: Analysing the Effects of Coupling Nebulization to Noninvasive Ventilation Through Pulmonary Scintigraphy on the Radioaerosol Deposition During Asthma Exacerbation
Brief Title: Radioaerosol Pulmonary Deposition During Asthma Exacerbation Through Noninvasive Ventilation
Acronym: NV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Valdecir Castor Galindo Filho, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: VNI1972NEB
Record Dates: First submitted 2009-04-22; First posted 2009-11-11 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Asthma
Keywords: Asthma; status asthmatics
MeSH Terms: conditions — Asthma | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NV Group (Experimental): Performed nebulization coupled with noninvasive ventilation
  Interventions: Device: NV
- NEB group (Active Comparator): Performed nebulization alone.
  Interventions: Other: NEB group

INTERVENTIONS:
Device: NV — Noninvasive ventilation coupled with nebulization(Nebulization containing salbutamol (2.5mg) and ipratropium bromide (0.25mg)plus oxygen flow in 7Lpm)
  Other Names: Interventional Group
  Arms: NV Group
Other: NEB group — Nebulization containing salbutamol (2.5mg) and ipratropium bromide (0.25mg)plus oxygen flow in 7Lpm
  Other Names: Control group
  Arms: NEB group

SUMMARY:
Despite the physiologic and clinical effects provided by coupling nebulization with noninvasive ventilation in asthma exacerbation, there are few and controversial studies reported in the literature.

DETAILED DESCRIPTION:
Reduced work of breathing, increased oxygenation and increased in expiratory peak flow (EPF) and forced expiratory volume in the first second (FEV1) are benefits of noninvasive ventilation (NV) in the treatment of asthma. Despite these clinical improvements attributed to NV during asthma exacerbations and the well-established effects of nebulization, there are few studies in the literature coupling both therapeutic resources.

In addition to this, no studies on scintigraphic analysis of radioaerosol deposition coupled with NV in asthmatics have published. A previous study was published by our group, but involved healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe asthma (FEV1 < 60 % of predicted values)
* Breathing rate > 25 bpm
* History of asthma for at least 1 year
* Duration of current asthma attack of < 7 days
* Reversibility of FEV1 of at least ≤ 10% after the administration of bronchodilator drugs

Exclusion Criteria:

* Current smoker
* Presence of cardiopulmonary disease (COPD, pneumonia, heart failure, myocardial infarction, pneumothorax)
* Hyperthermia
* Indication of intubation and invasive mechanical ventilation;
* Hemodynamic instability (heart rate > 150 bpm and systolic blood pressure < 90 mmHg)
* Cardiac arrhythmia
* Changes in consciousness
* Pregnancy
* Contraindications to use NV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary characteristics | 6 months

SECONDARY OUTCOMES:
Radioaerosol pulmonary index, radioaerosol penetration index and pulmonary clearance. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Valdecir C Galindo, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Valdecir Castor Galindo Filho, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Soroksky A, Stav D, Shpirer I. A pilot prospective, randomized, placebo-controlled trial of bilevel positive airway pressure in acute asthmatic attack. Chest. 2003 Apr;123(4):1018-25. doi: 10.1378/chest.123.4.1018. PMID 12684289
- [Background] Franca EE, Dornelas de Andrade AF, Cabral G, Almeida Filho P, Silva KC, Galindo Filho VC, Marinho PE, Lemos A, Parreira VF. Nebulization associated with bi-level noninvasive ventilation: analysis of pulmonary radioaerosol deposition. Respir Med. 2006 Apr;100(4):721-8. doi: 10.1016/j.rmed.2005.07.012. Epub 2005 Aug 31. PMID 16139491
- [Background] Soma T, Hino M, Kida K, Kudoh S. A prospective and randomized study for improvement of acute asthma by non-invasive positive pressure ventilation (NPPV). Intern Med. 2008;47(6):493-501. doi: 10.2169/internalmedicine.47.0429. Epub 2008 Mar 17. PMID 18344635
- [Derived] Galindo-Filho VC, Brandao DC, Ferreira Rde C, Menezes MJ, Almeida-Filho P, Parreira VF, Silva TN, Rodrigues-Machado Mda G, Dean E, Dornelas de Andrade A. Noninvasive ventilation coupled with nebulization during asthma crises: a randomized controlled trial. Respir Care. 2013 Feb;58(2):241-9. doi: 10.4187/respcare.01371. PMID 22781558
- See also: Related Info — http://www.nlm.nih.gov/medlineplus/asthma.html
- See also: Related Info — http://www.asthma.org.uk/